CLINICAL TRIAL: NCT02001363
Title: Protective Effect of Glucagonlike Peptide-1 on Reperfusion Injury in Patients With Acute Myocardial Infarction
Brief Title: Efficacy Study of Glucagonlike Peptide-1 to Treat Reperfusion Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chen Wei Ren, MD (Other)
Responsible Party: Sponsor-Investigator, Chen Wei Ren, MD, Dr., Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S2013-099-01; ChinaPLAGH (Other: ChinaPLAGH)
Record Dates: First submitted 2013-11-27; First posted 2013-12-04 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Acute Myocardial Infarction
Keywords: Reperfusion injury; Liraglutide
MeSH Terms: conditions — Reperfusion Injury | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- liraglutide (Experimental): drug: liraglutide (Novo Nordisk, Bagsværd, Denmark) duration:7 days(from admission (primary percutaneous coronary intervention) to discharge) the intervention:once-daily subcutaneous liraglutide 0.6 mg for 2 days, then gradually increase the dosage, once-daily subcutaneous liraglutide 1.2 mg for 2 days ,once-daily subcutaneous liraglutide 1.8 mg for 3 days
  Interventions: Drug: liraglutide (Novo Nordisk, Bagsværd, Denmark)
- liraglutide placebo (Placebo Comparator): drug:liraglutide placebo (Novo Nordisk) duration:7 days(from admission (primary percutaneous coronary intervention) to discharge) the intervention:once-daily subcutaneous liraglutide placebo 0.6 mg for 2 days, then gradually increase the dosage, once-daily subcutaneous liraglutide placebo 1.2 mg for 2 days ,once-daily subcutaneous liraglutide placebo 1.8 mg for 3 days
  Interventions: Drug: liraglutide placebo (Novo Nordisk)

INTERVENTIONS:
Drug: liraglutide (Novo Nordisk, Bagsværd, Denmark) — once-daily subcutaneous liraglutide 0.6 mg for 2 days, then gradually increase the dosage, once-daily subcutaneous liraglutide 1.2 mg for 2 days ,once-daily subcutaneous liraglutide 1.8 mg for 3 days
  Arms: liraglutide
Drug: liraglutide placebo (Novo Nordisk) — once-daily subcutaneous liraglutide placebo 0.6 mg for 2 days, then gradually increase the dosage, once-daily subcutaneous liraglutide placebo 1.2 mg for 2 days ,once-daily subcutaneous liraglutide placebo 1.8 mg for 3 days
  Arms: liraglutide placebo

SUMMARY:
The investigators planned to research the cardioprotective effects of intravenous liraglutide on reperfusion injury.

DETAILED DESCRIPTION:
Acute myocardial infarction is a major cause of mortality and morbidity. Primary percutaneous coronary intervention (pPCI) is currently the most effective treatment strategy in acute myocardial infarction. However, a sizable number of patients fail to restore optimal myocardial reperfusion, mostly because of the 'no-reflow' phenomenon. Glucagon-like peptide-1 (GLP-1) is an incretin hormone that regulates plasma glucose, and recently GLP-1 analogues have been introduced for the treatment of type-2 diabetes. In experimental studies, GLP-1 or its analogues protect against reperfusion injury-induced cell death. Exenatide reduces reperfusion injury in patients with ST-segment elevation myocardial infarction. Liraglutide(GLP-1) is safe and effective to reduce weight,serum lipid levels and blood pressure. Liraglutide can reduce cardiac rupture (12 of 60 versus 46 of 60; P=0.0001) and infarct size (21±2% versus 29±3%, P=0.02) and improved cardiac output (12.4±0.6 versus 9.7±0.6 ml/min; P=0.002) in normal and diabetic mice. The investigators planned to research the cardioprotective effects of intravenous liraglutide administered prior to reperfusion and continued after restoration of coronary blood flow in patients with STEMI undergoing pPCI.

ELIGIBILITY:
Inclusion Criteria:

Patients were eligible if they were 18 years or older and presented within 12 h from the onset of symptoms and signs of ST-segment elevation myocardial infarction to the catheterization laboratory.

Exclusion Criteria:

The patients were not considered for enrolment if they presented with unconsciousness, cardiogenic shock, hypoglycaemia, diabetic ketoacidosis, previous myocardial infarction, stent thrombosis, known renal insufficiency, or previous coronary artery bypass operation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
the salvage index measured by cardiac magnetic resonance | 3 months after primary percutaneous coronary intervention
  The primary endpoint was the salvage index measured by cardiac magnetic resonance after 3 months.

SECONDARY OUTCOMES:
major adverse cardiovascular events (MACE) after 3 months | 3 months after Primary percutaneous coronary intervention
  major adverse cardiovascular events (MACE) after 3 months: recurrent myocardial infarction, recurrent angina, revascularization, heart failure, cardiac death.
  treatment-emergent adverse events (TEAEs): hypoglycemia, nausea, acute pancreatitis
final infarct size after 3 months | 3 months after Primary percutaneous coronary intervention
the levels of high-sensitivity C-reactive protein (hsCRP) | 3 months after Primary percutaneous coronary intervention
nitric oxide (NO) levels | 3 months after Primary percutaneous coronary intervention

CONTACTS AND LOCATIONS:
Overall Officials: Yun Dai Chen, M.D., Study Director — World Health Organization
Locations (1):
- PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Garber A, Henry R, Ratner R, Garcia-Hernandez PA, Rodriguez-Pattzi H, Olvera-Alvarez I, Hale PM, Zdravkovic M, Bode B; LEAD-3 (Mono) Study Group. Liraglutide versus glimepiride monotherapy for type 2 diabetes (LEAD-3 Mono): a randomised, 52-week, phase III, double-blind, parallel-treatment trial. Lancet. 2009 Feb 7;373(9662):473-81. doi: 10.1016/S0140-6736(08)61246-5. Epub 2008 Sep 24. PMID 18819705
- [Background] Lonborg J, Vejlstrup N, Kelbaek H, Botker HE, Kim WY, Mathiasen AB, Jorgensen E, Helqvist S, Saunamaki K, Clemmensen P, Holmvang L, Thuesen L, Krusell LR, Jensen JS, Kober L, Treiman M, Holst JJ, Engstrom T. Exenatide reduces reperfusion injury in patients with ST-segment elevation myocardial infarction. Eur Heart J. 2012 Jun;33(12):1491-9. doi: 10.1093/eurheartj/ehr309. Epub 2011 Sep 14. PMID 21920963
- [Background] Liu H, Dear AE, Knudsen LB, Simpson RW. A long-acting glucagon-like peptide-1 analogue attenuates induction of plasminogen activator inhibitor type-1 and vascular adhesion molecules. J Endocrinol. 2009 Apr;201(1):59-66. doi: 10.1677/JOE-08-0468. Epub 2009 Jan 9. PMID 19136619
- [Result] Noyan-Ashraf MH, Momen MA, Ban K, Sadi AM, Zhou YQ, Riazi AM, Baggio LL, Henkelman RM, Husain M, Drucker DJ. GLP-1R agonist liraglutide activates cytoprotective pathways and improves outcomes after experimental myocardial infarction in mice. Diabetes. 2009 Apr;58(4):975-83. doi: 10.2337/db08-1193. Epub 2009 Jan 16. PMID 19151200
- [Derived] Huang M, Wei R, Wang Y, Su T, Li Q, Yang X, Chen X. Protective effect of glucagon-like peptide-1 agents on reperfusion injury for acute myocardial infarction: a meta-analysis of randomized controlled trials. Ann Med. 2017 Nov;49(7):552-561. doi: 10.1080/07853890.2017.1306653. Epub 2017 Mar 31. PMID 28286967
- [Derived] Chen WR, Chen YD, Tian F, Yang N, Cheng LQ, Hu SY, Wang J, Yang JJ, Wang SF, Gu XF. Effects of Liraglutide on Reperfusion Injury in Patients With ST-Segment-Elevation Myocardial Infarction. Circ Cardiovasc Imaging. 2016 Dec;9(12):e005146. doi: 10.1161/CIRCIMAGING.116.005146. PMID 27940956